CLINICAL TRIAL: NCT03134755
Title: Stress and Treatment Response in Puerto Rican Children With Asthma
Acronym: STAR
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan Celedon, MD, Professor, University of Pittsburgh
Other Study IDs: PRO17030493; R01HL117191 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Asthma in Children
Keywords: Asthma; Children; Stress; Puerto Rican; Health disparities; Treatment response; African American
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal epithelial samples for DNA and RNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort (all children with asthma): 300 children with asthma will receive the same inhaled corticosteroid (ICS) for six weeks, in order to assess response to ICS.Bronchodilator response will be measured before and after ICS therapy. Stress levels (the exposure of interest) will be assessed with a validated questionnaire, before ICS administration (thus, it is an observational study of whether stress is related to treatment response)
  Interventions: Drug: Inhaled corticosteroid (mometasone)

INTERVENTIONS:
Drug: Inhaled corticosteroid (mometasone) — The investigators are not measuring the effect of the intervention (ICS), but rather the effect of stress (which is not being intervened on), and this is thus an observational study. The ICS is given to children with asthma in whom an ICS is clinically indicated
  Other Names: Asmanex

SUMMARY:
This study aims to first determine whether high child stress leads to reduced response to common treatmenIs for asthma (inhaled corticosteroids and short-acting bronchodilators), and then to identify DNA methylation differences leading to stress-induced treatment resistance among children with asthma.

DETAILED DESCRIPTION:
Puerto Rican (PR) and African American children share a disproportionate burden from asthma in the U.S. The investigators have demonstrated that in PR children, a variety of psychological stressors are associated with worse asthma outcomes. Puerto Rican children also have reduced response to bronchodilators (short-acting inhaled β2-agonists, the most commonly used medication for asthma worldwide). The investigators have recently shown that high child stress is associated with reduced response to short-acting inhaled β2-agonists (bronchodilator response or BDR) in PR and non-PR children with asthma, and our preliminary results also implicate genetic and epigenetic (DNA methylation) variation in genes involved in stress responses (e.g., ADCYAP1R1) on asthma and BDR. Moreover, external in vitro experiments show that high stress leads to reduced expression of the genes for the β2-adrenergic receptor (ADRB2) and the glucocorticoid receptor (NR3C1) in white blood cells of children with asthma. While it is known that stress reduces BDR, it is not known whether this can be prevented by treatment with inhaled corticosteroids (ICS), or whether stress reduces response to ICS in vivo. Moreover, the research community has very limited knowledge of the genetic or epigenetic mechanisms underlying treatment resistance in stressed children. On the basis of novel preliminary results, the investigators hypothesize that chronic stress reduces response to inhaled corticosteroids (ICS) and BDR in PR and African American children with asthma, and that these effects are mediated by altered methylation of genes regulating responses to stress, corticosteroids and BDR. To test this hypothesis, the investigators will first determine whether increased stress leads to reduced response to ICS or BDR (even after treatment with ICS) in 300 PR and African American children with asthma (Aim 1). The investigators will then test for association between high child stress and genome-wide DNA methylation in respiratory (nasal) epithelium in 550 Puerto Rican and African American children with asthma (Aim 2). Next, the investigators will examine whether methylation changes in the top 100 genes identified in Aim 2 are associated with response to ICS or BDR in 300 to 550 PR and African American children with asthma (Aim 3a). Finally, the investigators will assess the effects of methylation changes identified in Aim 3a on gene expression (Aim 3b). This proposal should determine whether and how psychosocial stress leads to reduced response to common treatments for asthma control (ICS) and relief of asthma symptoms (short-acting inhaled β2-agonists) in a high-risk group (Puerto Rican and African American children).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* BDR ≥8%99 or (if BDR<8%) increased airway responsiveness to methacholine (PD20 <16.81 umol)
* Four Puerto Rican grandparents
* Steroid naïve (no treatment with ICS, nasal, or oral corticosteroids in the prior 4 weeks)
* Parental consent and child's assent to participate in the study

Exclusion Criteria:

* Chronic disease (i.e. respiratory, liver, cardiac, renal, neurologic) other than asthma
* Severe asthma, as evidenced by: a) intubation for asthma at any time, or b) ≥3 hospitalizations or ≥6 visits to the emergency department/urgent care in the previous year, or c) chronic/continuous need for medications other than single controller therapy [ICS or leukotriene inhibitors] and short-acting β2-agonists
* Current smoking or former smoking if ≥5 pack-years
* Inability to perform acceptable spirometry
* FEV1 <60% of predicted

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 300 Puerto Rican and African American children with mild to moderate persistent asthma, ages 8 to 20 years. Of these children, 150 (all Puerto Rican) will be recruited in the metropolitan area of San Juan and Caguas (Puerto Rico), and 150 (all African American) will be recruited in Pittsburgh (PA).
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Bronchodilator response (BDR) | 15 minutes
  BDR will be measured as the change in forced expiratory volume in 1 second (FEV1) after administration of a short-acting bronchodilator (albuterol)
Response to inhaled corticosteroids (ICS) | Six weeks
  ICS response will be measured as change in forced expiratory volume in 1 second (FEV1) and as change in the xhild-Asthma Control Test (C-ACT) score, following six weeks of ICS administration
DNA methylation and gene expression differences | Six weeks
  The investigators will examine whether child stress is associated with DNA methylation or gene expression differences, and such differences will then be tested for association with BDR or ICS response (measured as above)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Celedon, MD, DrPH, Principal Investigator — University of Pittsburgh
Locations (2):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States
- Behavioral Sciences Research Institute, University of Puerto Rico, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No